CLINICAL TRIAL: NCT05974449
Title: A Phase II Clinical Study of Lactobacillus Vaginalis Capsules for the Prevention and Treatment of Symptoms of Vulvovaginal Atrophy in Young Breast Cancer Patients Receving Ovarian Function Suppression (OFS) During Chemotherapy
Brief Title: Lactobacillus Vaginalis Capsules for Treatment of Vulvovaginal Atrophy in Young Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jue Wang, Prof., The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: BC-OFSAE-Lactobacillus
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Female
Keywords: Breast cancer, Vulvovaginal symptoms ，Lactobacillus capsules
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- C1, C2 dosing group (Experimental): C1 and C2 dosing groups: The drug is administered on the day of the C1 and C2 chemotherapy cycles for 10 days, washing the vulva and placing the drug deep into the vagina, once a night, 1 capsules each time.
  Interventions: Drug: Vaginal Lactobacillus capsules
- C3, C4 dosing group (Experimental): C3 and C4 dosing groups: The drug is given on the day of the C3 and C4 chemotherapy cycles and is administered for 10 days. The drug is placed deep into the vagina after washing the vulva, once a night, 1 capsules each time.
  Interventions: Drug: Vaginal Lactobacillus capsules

INTERVENTIONS:
Drug: Vaginal Lactobacillus capsules — This product is a micro-ecological preparation made from live Lactobacillus and is used for the treatment of vaginosis caused by disorders of the flora.
  Other Names: Ding Jun Sheng

SUMMARY:
This study is a prospective, randomized controlled, phase II clinical study with a planned enrolment of 60 patients. The study focuses on the efficacy and safety of Lactobacillus vaginalis capsules for the prevention and/or treatment of vulvovaginal symptoms in young breast cancer patients receiving ovarian protection during chemotherapy, in order to improve compliance and quality of life in breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women, and its incidence is increasing year by year. While systemic combination therapy (e.g., Chemotherapy, endocrine therapy, targeted therapy, etc.) can increase the cure rate of patients, it can also bring about some adverse effects that can negatively affect the life of patients. The most common form of chemotherapy, for example, is chemotherapy drugs (especially cyclophosphamide-containing chemotherapy regimens), which can lead to impaired ovarian function. Inhibition of ovarian function with gonadotropin-releasing hormone agonists (GnRHa) can achieve protection of the ovaries during chemotherapy and help restore ovarian function. As the trend towards younger breast cancer has become more pronounced in recent years, ovarian protection has also received increasing attention. However, ovarian protection can also dramatically reduce serum estrogen levels in patients, leading to vulvovaginal symptoms such as vaginal dryness, difficulty with intercourse, genital skin irritation, itching, burning, and increased vaginal discharge. Moreover, patients are often too shy to express these symptoms, leading to underdiagnosis and under-treatment.

The North American Menopause Society states that topical estrogen therapy is the first-line option for moderate to severe vulvovaginal symptoms, but its safety in women with breast cancer is not known. Some studies have shown an increase in serum estradiol levels with the use of estradiol vaginal rings and creams, and there are no clinical studies to suggest a relationship between a mild increase and the risk of breast cancer recurrence. and short-term effects are limited. --The hierarchy is not out: hormonal therapy first, then non-hormonal therapy The onset of vulvovaginal symptoms is primarily due to a decrease in serum circulating estrogen in women, but many researchers are beginning to explore whether these changes can be attributed to changes in the dynamics of the vaginal microbiome. The vaginal microecology of healthy women is dominated by lactic acid bacteria, which proliferate in the anaerobic environment of the vagina, producing various antimicrobial compounds such as lactic acid, hydrogen peroxide (H2O2) and bacteriocins and maintaining vaginal health by enhancing epithelial barrier function, symbiotic colonization, blocking pathogenic bacterial adhesion, lowering pH, influencing antimicrobial peptide production/secretion and overall mucosal immunity. In patients presenting with vulvovaginal symptoms, vaginal microecology is no longer dominated by lactobacilli and it has been shown that the severity of vaginal dryness, dyspareunia, and vaginal pain symptoms are negatively correlated with the number of lactobacilli in the vagina. To address this issue, researchers have explored the fact that Donders et al. found that Lactobacillus combined with low-dose estrogen significantly improved vulvovaginal symptoms in women but caused a concomitant increase in serum estradiol, the risk of which is not yet known in breast cancer patients , whereas this study explored the use of Lactobacillus alone as an intervention to see if there was an increase in serum estradiol after the intervention, and prophylactic medication was administered to address patients who endure vulvovaginal symptoms due to shyness of expression. However, there is a lack of large randomized controlled clinical studies to determine the effectiveness of Lactobacillus in modulating or restoring a dysregulated vaginal microbiome and improving vaginal symptoms in different populations. The aim of this study was to explore, in the small sample size, whether prophylactic use of Lactobacillus vaginalis capsules during ovarian protection in breast cancer patients could prevent vulvovaginal symptoms in patients and to assess its safety in order to improve treatment adherence in breast cancer patients and improve the quality of life of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed invasive breast cancer (regardless of pathology type);
2. Female patients 18-40 years of age with unlimited HR, or 41-45 years of age with negative HR;
3. Patients expected to receive ≥4 cycles of chemotherapy containing paclitaxel or anthracycline-containing chemotherapeutic agents and ovarian protective drugs;
4. Pre-menopausal (including perimenopausal);
5. Good compliance, normal comprehension and ability to receive treatment as required;
6. ECOG score 0-1;
7. Patients volunteered to participate in this study and signed an informed consent form.

Exclusion Criteria:

1. Use of any other vaginal medication in the 3 months prior to the study;
2. Use of any anti-infective medication in the 3 months prior to the study;
3. Active genital tract infection;
4. Previous development of other malignancies;
5. Any reason why they are unable to complete the full course of follow-up treatment as prescribed by their doctors;
6. AST and ALT ≥ 1.5 times the upper limit of normal, alkaline phosphatase ≥ 2.5 times the upper limit of normal, total bilirubin ≥ 1.5 times the upper limit of normal, serum creatinine ≥ 1.5 times the upper limit of normal; LVEF < 50% on cardiac ultrasound;
7. Severe coagulation disorder, severe systemic disease, or uncontrollable infection;
8. Persons without personal freedom and independent civil capacity; the presence of mental disorders, addictions, etc., which in the judgment of the investigator do not qualify for enrolment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal PH | 1 year
  Reactive vaginal pH
Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) | 1year
  For assessing quality of life and vulvovaginal symptoms in women. Using "Absolutely not", "A little", "Some", "Very", "Extremely" to indicate the severity of symptoms

SECONDARY OUTCOMES:
The detection rate of vaginal secretions of Gardnerella vaginalis, Lactobacillus janus, Lactobacillus garciae, Lactobacillus curvatus, Lactobacillus inertus, Lactobacillus chimaerae, Prevotella spp. and Streptococcus spp; | 1year
  Detection of target flora in vaginal secretions using qPCR. Reflecting changes in vaginal microecology.
Serum concentrations of estrone, estradiol and oestrogen binding protein | 1 year
  Testing serum hormone levels

CONTACTS AND LOCATIONS:
Overall Officials: Jue Wang, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No